CLINICAL TRIAL: NCT03329261
Title: Incidence Des évènements cArdiovasculaires majeurS Chez Les Patients COronariens diabétiques Subissant Une angioPlastie Coronaire et traités Par Clopidogrel à la Dose 150 mg Versus 75 mg
Brief Title: Incidence of Major Cardiovascular Events in Diabetic Patients With ACS Undergoing Coronary Angioplasty and Treated With Clopidogrel 150 mg Versus 75 mg
Acronym: IDASCOP 1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoires Teriak (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERIAK-001
Record Dates: First submitted 2017-10-14; First posted 2017-11-01 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Diabetes Mellitus, Type 2; NSTEMI - Non-ST Segment Elevation MI; Coronary Angioplasty
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-ST Elevated Myocardial Infarction | interventions — Clopidogrel

STUDY DESIGN:
Intervention Model Description: A comparative, interventional, multicenter, randomized, prospective, two-arm study with monotherapy in two different doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (single dose) (Active Comparator): Will receive a clopidogrel loading dose of 600 mg PO, then a daily dose of clopidogrel 75 mg PO until the angioplasty is performed. After coronary intervention, a daily dose of clopidogrel 150 mg PO for 7 days will be given, followed by a daily single dose of clopidogrel (75 mg PO) for 21 days. Maintenance therapy will be clopidogrel daily dose of 75 mg PO thereafter, until the end of the study.
  Interventions: Drug: Clopidogrel
- Arm 2 (double dose) (Active Comparator): Will receive a clopidogrel loading dose of 600 mg PO, then a daily dose of clopidogrel 75 mg PO until the angioplasty is performed. After coronary intervention, a daily dose of clopidogrel 150 mg PO for 7 days will be given, followed by a daily double dose of clopidogrel (150 mg PO) for 21 days. Maintenance therapy will be clopidogrel daily dose of 75 mg PO thereafter, until the end of the study.
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Clopidogrel — COPIGREL® - clopidogrel dosed at 75 mg per tablet
  Other Names: COPIGREL®

SUMMARY:
Acute Coronary Syndrome (ACS) is triggered by the rupture of an atherosclerotic plaque that results in a platelet aggregation reaction in the coronary artery. The administration of antiplatelet agents starting from the acute phase of the disease has helped reduce the risk of ischemic relapse both during initial and long-term hospitalization.

Management of clopidogrel following an ischemic event has been the subject of several treatment regimens ranging from a single continuous dose to a sequential double dose of between 7 and 30 days. The CURRENT-OASIS 7 therapeutic trial showed a benefit of clopidogrel double dose in reducing the risk of myocardial intervention (MI) and the composite outcome: cardiovascular mortality, MI, or stroke (CVA/TIA) at 30 days. However, the study protocol was interested in all ACSs, regardless of the Type 2 Diabetes Mellitus (T2DM) status in selected patients. Also, doubling of clopidogrel dose was maintained over 7 days after angioplasty. The literature describes an increased cardiovascular risk in type II diabetics in secondary prevention. No previous study has evaluated the effect of clopidogrel double dose given for 1 month on the reduction of this risk in the long-term in diabetic patients.

Thus, the objective of this study is to evaluate the efficacy and safety of clopidogrel double dose, given for 1 month in ACS in the diabetic patient.

DETAILED DESCRIPTION:
The study is an open label, multicentric clinical trial. Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion criteria:

* Male or female aged between 18 to 75 years old.
* Proven ACS requiring PTCA within 1 week of inclusion. The ACS should be without ST-segment elevation (presence of chest pain with ST-segment or T-wave changes without sustained ST segment elevation) with elevation of cardiac biomarkers of MI (positive troponins).
* Coronary angiography showing at least one coronary lesion, whether mono, bi or multi-truncate
* Type 2 diabetes confirmed for at least one year
* Patient candidate for treatment with Clopidogrel
* Informed consent of patients

Non-Inclusion Criteria:

* Non-consenting patient and/or participating in another clinical study
* ACS with ST segment elevation (STEMI)
* History of digestive or cerebral bleeding with antiplatelet agents or anticoagulants
* Insulin-dependent diabetes mellitus (IDDM)
* Diabetic requiring insulin
* Patient in cardiogenic shock
* Patient under treatment with anti-glycoprotein IIb/IIIa or stopped less than 72 hours prior to inclusion
* Previously treated with clopidogrel or thrombolytics
* Patients programmed for surgery in less than 6 months
* Ischemic stroke less than 6 weeks old
* History of haemorrhagic stroke (regardless of time)
* Patients under or candidates for Vitamin K antagonist (VKA)
* Patients under another antiplatelet agent (Ticlopidine, Prasugrel)
* Patients with a contraindication to clopidogrel (hypersensitivity to the active substance or to any of the excipients, severe hepatic impairment, progressive hemorrhagic lesion such as peptic ulcer or intracranial hemorrhage)
* Under omeprazole treatment, or considered during the study
* Anemia (Hb <12g/dl)
* Thrombocytopenia with less than 100000 cells/mm3
* Serum creatinine greater than 200 μmol/l
* Pregnancy and/or breast-feeding
* Severe renal impairment

Exclusion criteria:

* Non-compliance with treatment (treatment compliance <80%)
* AE/SAE requiring cessation of treatment
* Planning a CABG
* Occurrence of pregnancy during the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-03-24 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Major Cardiovascular Events (MACE) | 1 year after coronary intervention
  Incidence of major cardiovascular events including cardiac death, MI, cerebrovascular accident (CVA), revascularization (PTCA, GABG), stent thrombosis.

SECONDARY OUTCOMES:
Bleeding Events | At 1, 3, 6, 9 and 12 months from patient enrollment
  All bleeding events (digestive, cerebral, other locations)
Heart Failure Readmission | At 1, 3, 6, 9 and 12 months from patient enrollment
  Incidence of heart failure hospital readmissions
Global Death | At 1, 3, 6, 9 and 12 months from patient enrollment
  Incidence of death of all causes (death of cardiovascular origin and death of non-cardiovascular origin)
Incidence of Adverse Events | At 1, 3, 6, 9 and 12 months from patient enrollment
  Incidence of Adverse Events (AE) including Serious Adverse Events (SAE)

CONTACTS AND LOCATIONS:
Locations (1):
- HMPIT, Ben Arous, Tunisia